CLINICAL TRIAL: NCT00247221
Title: Family Motivational Interviews for ETOH+ Teens in the ER
Brief Title: Brief Intervention for Families of Teens Treated in the Emergency Department for an Alcohol-Related Event
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAASPI013385; R01AA013385 (NIH); NIH grant R01 AA013385
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Alcohol Abuse
Keywords: Alcohol; Substance abuse; Adolescent; Family functioning
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1) MI/Family Check-Up (Experimental): Brief integrated individual and family intervention -- the experimental intervention integrates an individual Motivational Interview (MI) for the adolescent with a brief family intervention, the Family Check-Up
  Interventions: Behavioral: MI/Family Check-up
- 2) MI only (Active Comparator)
  Interventions: Behavioral: MI only

INTERVENTIONS:
Behavioral: MI/Family Check-up — The experimental intervention integrates an individual Motivational Interview (MI) for the adolescent with a brief family intervention, the Family Check-Up. Follow-up interviews will be conducted at 3, 6, and 12 months after the baseline intervention.
  Arms: 1) MI/Family Check-Up
Behavioral: MI only — An individual motivational interview (IMI only) will be conducted at 3, 6, and 12 months after the baseline intervention to assess outcome.
  Arms: 2) MI only

SUMMARY:
The purpose of this study is to compare the effectiveness of a brief family intervention in reducing alcohol use and alcohol-related problems among families of underage drinkers (13-17 years old) who are treated in a hospital emergency department for an alcohol-related event.

DETAILED DESCRIPTION:
The long-term objectives of this research program are to develop effective interventions in health care settings for reducing problem drinking and associated problems among adolescents and to further enhance intervention approaches by identifying effective elements of treatment. The major purpose of this study is to compare a brief integrated individual and family intervention designed to reduce alcohol use and related problems to an enhanced standard care condition (standard care plus family assessment).

The targeted population is underage drinkers (13-17 years old) who have been treated in an Emergency Department following an alcohol-related event. It is important to intervene with this population because alcohol-involved adolescents may be at higher risk for having continuing alcohol problems (Fillmore, 1988; Zucker, in press). The intervention is conceptualized as using a "teachable moment" (i.e., shortly after a salient event) to increase family interest in reducing harmful drinking. The experimental intervention integrates an individual Motivational Interview (MI) for the adolescent, based on our research group's prior work with this intervention, with a brief family intervention, the Family Check-Up (Dishion & Kavanagh, 2003).

The experimental condition will be compared to standard care plus family assessment. This design allows us to test the added benefit of the brief family intervention compared to the benefits often derived from assessment without added treatment. Follow-up interviews will be conducted at 3, 6, and 12 months after the baseline intervention to assess outcome. The specific aims of this proposal are to test the effectiveness of the experimental intervention in reducing alcohol-related problems, alcohol consumption, and other behavior problems compared to the enhanced standard care condition. Second, we will examine whether depressed mood and behavior problems at baseline moderate the effects of the treatment conditions. We will also test whether individual factors (motivation to change behavior) and environmental factors (parent/family influence and peer influence) mediate the relation between the treatment condition and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 13-17 years
* Receiving treatment at the approved medical Emergency Department
* Child living in a home with at least one parent or legal guardian

Exclusion Criteria:

* Children who are suicidal, in police custody, not alert/oriented, non-English speaking, in severe pain, or who have sustained severe trauma
* Children with a history of prior substance abuse treatment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2002-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Alcohol use | 3 months
  Drinking frequency (days per month), quantity (drinks per occasion), and frequency of high-volume drinking (5 or more drinks per occasion) over the prior 3 months.
Alcohol use | 6 months
  Drinking frequency (days per month), quantity (drinks per occasion), and frequency of high-volume drinking (5 or more drinks per occasion) over the prior 3 months.
Alcohol use | 12 months
  Drinking frequency (days per month), quantity (drinks per occasion), and frequency of high-volume drinking (5 or more drinks per occasion) over the prior 3 months.

SECONDARY OUTCOMES:
marijuana use | 3 months
  Days of use in prior 3 months
Marijuana use | 6 months
  Days of use in prior 3 months
Marijuana use | 12 months
  Days of use in prior 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Study Director — Brown University
Locations (1):
- Rhode Island Hospital/Lifespan Corporation and Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Spirito A, Sindelar-Manning H, Colby SM, Barnett NP, Lewander W, Rohsenow DJ, Monti PM. Individual and family motivational interventions for alcohol-positive adolescents treated in an emergency department: results of a randomized clinical trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):269-74. doi: 10.1001/archpediatrics.2010.296. PMID 21383276